CLINICAL TRIAL: NCT06967298
Title: How Does Total 30 Sphere Perform in Those Who Previously Dropped Out of Contact Lenses Due to Comfort or Dryness?
Brief Title: Total30 For Contact Lens Dropouts
Acronym: T30DO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern College of Optometry (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: irb00006763
Record Dates: First submitted 2025-02-21; First posted 2025-05-13 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye; Contact Lens Complication; Contact Lenses
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: This prospective 6 month 4 visit survey will refit individuals who have previously dropped out of contact lenses that is stopped wearing them due to discomfort into T30 contact lenses to determine if they are comfortable.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- T30 For Dropouts (Experimental): Total 30 contact lenses for those who have previously dropped out of CL wear
  Interventions: Device: T30 Contact lenses

INTERVENTIONS:
Device: T30 Contact lenses — Individuals who have previously dropped out of Contact lenses (CL) due to discomfort will be refit into T30 contact lenses and their comfort with the product will be assessed.

SUMMARY:
Contact lens (CL) discomfort is a complex phenomenon that has been defined by the Tear Film and Ocular Surface Society (TFOS) in their seminal report on CL discomfort as a condition that results in "episodic or persistent adverse ocular sensation related to lens wear, either with or without visual disturbance resulting from reduced compatibility between the CL and the environment, which can lead to decreased wearing time and discontinuation of CL wear."

DETAILED DESCRIPTION:
Contact lens (CL) discomfort is a complex phenomenon that has been defined by the Tear Film and Ocular Surface Society (TFOS) in their seminal report on CL discomfort as a condition that results in "episodic or persistent adverse ocular sensation related to lens wear, either with or without visual disturbance resulting from reduced compatibility between the CL and the environment, which can lead to decreased wearing time and discontinuation of CL wear."1 While CL dropout occurs in about 20% of wearers annually the majority of CL wearers who cease wearing their CLs have a desire to continue wearing their CL if given the opportunity.3 A recent review by Pucker and Tichenor found that CL discomfort was the top reason for established CL wears to cease wearing CLs Therefore, providing CL dropouts with an alternative material, which may be more comfortable than their past CLs, could be a means for curbing CL dropout.

Our recent work found that when 60 participants who had previously dropped out of CLs were given the opportunity to be refit into Dailies TOTAL1® CLs that 100% of them were still wearing Dailies TOTAL1® at 1 month and 98% of them were still wearing their CLs at 6 months. When these participants were asked at the 1-month visit, 98.3%, 86.5%, and 93.2% of them responded that they were very satisfied or satisfied with their vision, their end-of-day CL comfort, and overall CL comfort, respectively. These same participants responded at 6 months that they were very likely or likely to continue to wear the study CLs (80.7%) and to recommend the study CLs to a friend (93.2%). While these data suggest that CL dropout can thrive when being refit into a daily disposable CLs, the literature currently lacks a targeted study aimed at understanding how CL dropouts will respond to being refit into a monthly replacement CL. One good potential monthly CL option is the TOTAL30® (T30) CL. T30 is a relatively new frequent replacement CL, with a biocompatible design. Thus, the purpose of this study is to determine the frequency that CL dropouts who dropped out of CLs because of dryness or discomfort can be comfortably refit into T30 CLs at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18- to 40-year-old, past CL wearers who have best corrected 20/20 visual acuity or better
* Participants will be required to have worn reusable CLs for at least one year in the past.
* Participants over the age of 40 years will be excluded to avoid presbyopia-related vision issues.
* Participants must have dropped out of reusable CLs within the past two years because of discomfort or dryness.

This determination will be made by listing Young et al.'s list of reasons for dropping out of CLs and asking the participants to indicate their top reason for dropping out of CLs:

a. Discomfort or Dryness b. General Poor Vision, c. Poor Reading Vision, d. Difficulty with Handling, e. Advised by Practitioner, f. Inconvenient, g. Eyes were Red, h. Lost Interest, i. Too Costly, j. Reaction to Care Products, k. Lost Lenses, l. Other.

* . Participants will be considered a CL dropout if they have not worn CLs in the past 3 months. Participants will be required to have scores of ≤3 on the SPEED questionaries' (no significant dry eye symptoms).
* Participants will be required to be able to wear T30 sphere CLs (astigmatism ≤ 0.75 D OD/OS).
* Participants will be required to provide a prescription for glasses that is less than 3 years old.

Exclusion Criteria:

* if they are past rigid CL wearers,
* have worn reusable CLs within the past two years,
* have a history of being diagnosed with dry eye or ocular allergies,
* have known systemic health conditions that are thought to alter tear film physiology,
* have a history of viral eye disease,
* have a history of ocular surgery,
* have a history of severe ocular trauma,
* have a history of corneal dystrophies or degenerations,
* have active ocular infection or inflammation,
* are currently using isotretinoin-derivatives or ocular medications, or
* if they are pregnant or breast feeding.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Likelihood of continuing to wear T30 CLs at 1 month and 6 months | 1 month and 6 months
  Participants will be refit into new contact lenses and their comfort will be asked about their comfort.In which a higher score is better.
Overall satisfaction while wearing T30 CLs at 1 month and 6 months. | 1-6 months
  Comfort in the lenses will be judged at 1 and 6 months to determine if the participant is satisfied using Visual Acuity scores in which higher scores are better.

CONTACTS AND LOCATIONS:
Locations (1):
- The Southern College of Optometry, Memphis, Tennessee, United States